CLINICAL TRIAL: NCT07144826
Title: A Randomized, Double-Blind, Placebo Controlled, Study to Investigate Efficacy of a Probiotic Intervention on the Gut and Vaginal Microbiome of Ovarian Cancer Patients Undergoing Treatment With Platinum Chemotherapy
Brief Title: Effects of a Probiotic Intervention on the Gut and Vaginal Microbiome in Patients With Advanced or Recurrent Ovarian Cancer Undergoing Treatment With Platinum Chemotherapy
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Laura Chambers, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OSU-24095; NCI-2025-05052 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Advanced Ovarian Carcinoma; Recurrent Ovarian Carcinoma; Stage II Ovarian Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Specimen Handling; Probiotics; Fluid Therapy; Powders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (probiotic) (Experimental): Patients receive probiotic PO BID beginning within seven days of SOC platinum chemotherapy cycle 1 until seven days after their cycle 6. Cycles repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood and vaginal sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Dietary Supplement: Probiotic; Other: Questionnaire Administration
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID beginning within seven days of SOC platinum chemotherapy cycle 1 until seven days after their cycle 6. Cycles repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood and vaginal sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and vaginal sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Placebo Administration — Given PO
  Arms: Arm II (placebo)
Dietary Supplement: Probiotic — Given PO
  Other Names: Probiotic Supplement; Probiotic supplements (pills, liquid, powder; or other probiotics)
  Arms: Arm I (probiotic)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the effects a probiotic intervention has on the gut and vaginal microbiome in patients undergoing chemotherapy for ovarian cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that has come back after a period of improvement (recurrent). Gut health is also known as the gut microbiome. The microbiome includes all of the bacteria and organisms naturally found in the digestive tract. Probiotics are dietary supplements containing live microorganisms that may help keep the gastrointestinal tract healthy. A probiotic intervention during platinum chemotherapy in ovarian cancer patients may impact the gut and vaginal microbiota, quality of life, symptoms, and oncologic outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate changes to the gut microbiome composition in ovarian cancer patients randomized to a probiotic intervention versus placebo during platinum chemotherapy.

SECONDARY OBJECTIVES:

I. Compliance with probiotic intervention in ovarian cancer patients during chemotherapy.

II. Compliance with gut microbiome collection in ovarian cancer patients during chemotherapy.

III. Compliance with vaginal microbiome collection in ovarian cancer patients during chemotherapy.

IV. Recurrence free survival (RFS). V. Overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To evaluate changes in the vaginal microbiome composition of ovarian cancer patients randomized to a probiotic intervention versus placebo during platinum chemotherapy.

II. Assess pre-chemotherapy diet according to the Food Frequency Questionnaire (FFQ, Diet History Questionnaire [DHQ3]) questionnaire and how this influences the patient's baseline gut and vaginal microbiome.

III. Assess whether a probiotic intervention influences chemotherapy toxicity and morbidity.

IV. Assess whether a probiotic intervention influences stool consistency or need for additional medications during chemotherapy.

V. Assess impact of gut and vaginal microbiome on patient quality of life. VI. Assess changes in serum metabolomic and immune markers as a result of the probiotic intervention.

VII. Assess whether probiotic intervention is associated with chemotherapy-induced neutropenia, neutropenic fever and dose-delays.

VIII. In patients who undergo standard-of-care surgery during chemotherapy, assessment of post-operative infectious outcomes, including surgical site infection in ovarian cancer patients randomized to a probiotic intervention versus placebo during platinum chemotherapy.

IX. In patients who undergo standard-of-care surgery during chemotherapy, assessment of the tumor microbiome as a result of probiotic intervention versus placebo.

X. In patients who are treated with antibiotics as standard of care for infectious causes during chemotherapy, assess changes in the vaginal and gut microbiome related to antibiotic therapy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive probiotic orally (PO) twice daily (BID) beginning within seven days of standard of care (SOC) platinum chemotherapy cycle 1 until seven days after their cycle 6. Cycles repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood and vaginal sample collection throughout the study.

ARM II: Patients receive placebo PO BID beginning within seven days of SOC platinum chemotherapy cycle 1 until seven days after their cycle 6. Cycles repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood and vaginal sample collection throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written consent form. In patients who do not speak English, ability to have informed consent form translated in their native language and have their native language translator present for consenting process
* Age > 18 years old
* Patient with advanced (stage II, III or IV) or recurrent ovarian cancer who will receive platinum-based chemotherapy as standard of care (cisplatin, carboplatin containing regimens)
* Agreeable to participate in all research activities defined in the study
* Agreeable to not take any other probiotic and/or prebiotic supplements outside of study intervention during the study
* Agreeable to not make significant changes to their diet throughout the course of the study
* Patients with ileostomy, colostomy are permitted to participate

Exclusion Criteria:

* Borderline ovarian tumors
* Prior allergy or food intolerance to any probiotic product
* History of chronic inflammation or active structural abnormality of the digestive tract (e.g., inflammatory bowel disease requiring medications, active duodenal or gastric ulcer, complete large or small bowel intestinal obstruction, active fistula)
* Patients who do not meet laboratory parameters for platinum-based chemotherapy, including absolute neutrophil count (ANC) < 1500
* Known hypersensitivity to any component of study product (Akkermansia muciniphila, Anaerobutyricum hallii, Clostridium beijerinckii, Clostridium butyricum and Bifidobacterium infantis, chicory inulin, magnesium stearate, grape food color, and silica)
* Known hypersensitivity to > 4 first-line antimicrobial therapies against Akkermansia muciniphila, Clostridium beijerinckii, Clostridium butyricum, Anaerobutyricum hallii: penicillin, piperacillin, tetracycline, amoxicillin, ampicillin
* Known hypersensitivity to > 4 first-line antimicrobial therapies against Bifidobacterium infantis Bi-26^Trademark (TM): gentamicin, kanamycin, streptomycin, tetracycline, erythromycin, clindamycin, ampicillin, vancomycin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Estimated)
Dates: Start 2026-01-09 (Estimated); Primary Completion 2027-07-09 (Estimated); Study Completion 2027-07-09 (Estimated)

PRIMARY OUTCOMES:
Changes to the gut microbiome composition | Within one week before or after cycle 1 of chemotherapy, within one week before or after cycle 3 of adjuvant chemotherapy, and within one week before or after cycle 6 of adjuvant chemotherapy (cycle length = 21 days)
  Will be assessed by stool samples collected from all patients. Microbe diversity and communities are assessed by 16s ribosomal ribonucleic acid sequencing and metagenomic whole-genome shotgun sequencing. Presence of microbes between responders and non-responders will be compared using Fisher's exact tests and logistic regression. Changes over time will be assessed using generalized linear or logistic regression models accounting for repeated measures, depending on the format of the outcome variable.

SECONDARY OUTCOMES:
Patient compliance with taking probiotic pills | At chemotherapy visits for cycle 2, 3, 4, 5, and 6 (cycle length = 21 days)
  Will be assessed by patient compliance with taking probiotic pills based on the number of pills dispensed versus number of pills remaining at visits, and reason for non-compliance. Compliance will be assessed with patient completion of surveys and return of kits by determining % of kits returned compared to those given to patients and assessing the period of time between when a microbiome kit was provided to a patient and when they returned it. All analyses will be done using SAS (version 9.4, The SAS Institute, Cary, North Carolina [NC]), and a p < 0.05 will be considered statistically significant.
Patient compliance with gut microbiome collection | Within one week before or after cycle 1 of chemotherapy, within one week before or after cycle 3 of adjuvant chemotherapy and within one week before or after cycle 6 of adjuvant chemotherapy (cycle length = 21 days)
  Will be assessed through number of stool sample kits returned to processing lab versus number of kits given out. Compliance will be assessed with patient completion of surveys and return of kits by determining % of kits returned compared to those given to patients and assessing the period of time between when a microbiome kit was provided to a patient and when they returned it. All analyses will be done using SAS (version 9.4, The SAS Institute, Cary, NC), and a p < 0.05 will be considered statistically significant.
Patient compliance with vaginal microbiome collection | Within one week before or after cycle 1 of chemotherapy, within one week before or after cycle 3 of adjuvant chemotherapy and within one week before or after cycle 6 of adjuvant chemotherapy (cycle length = 21 days)
  Will be assessed through number of vaginal microbiome swab sample kits returned to processing lab versus number of kits given out. Compliance will be assessed with patient completion of surveys and return of kits by determining % of kits returned compared to those given to patients and assessing the period of time between when a microbiome kit was provided to a patient and when they returned it. All analyses will be done using SAS (version 9.4, The SAS Institute, Cary, NC), and a p < 0.05 will be considered statistically significant.
Recurrence free survival (RFS) | Months from first cycle of chemotherapy (cycle 1) to time of recurrence defined by primary physician assessment (cycle length = 21 days)
  Kaplan Meier plots will be created to compare the RFS of patients treated with probiotic versus (vs.) placebo, and RFS will also be assessed based on the presence of specific gut microbes, with median RFS being reported, with 95% confidence intervals.
Overall survival (OS) | Months from first cycle of chemotherapy (cycle 1) to time of death (cycle length = 21 days)
  Kaplan Meier plots will be created to compare the OS of patients treated with probiotic vs. placebo, and OS will also be assessed based on the presence of specific gut microbes, with median OS times being reported, with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Chambers, DO, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu